CLINICAL TRIAL: NCT07191119
Title: Feasibility and Efficacy of Transcutaneous Auricular Vagus Nerve Stimulation for Insomnia in Survivors of Childhood Acute Lymphoblastic Leukemia
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation for Insomnia in Survivors of Childhood Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: FANSI
Record Dates: First submitted 2025-08-26; First posted 2025-09-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Survivor of Childhood Cancer; Insomnia; Acute Lymphoblastic Leukemia (ALL)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: A blinded, randomized sham/placebo-controlled pilot study with self-administered tVNS.
  While "Device Feasibility" generally has fewer than 10 participants, the aim is to ensure safety in a novel device population. While this does not fit into "Supportive Care," it also requires more participants for considerations:
  * Using a blinded 1:1 sham:verum study design with a control arm to ensure device feasibility is not affected by perceived stimulation. It is important to consider the inherent experience of tVNS.
  * As this is a novel population for the device and treatment, the study aims to ensure an adequate sample size to obtain effect size estimates to inform power analyses on future trials will be achieved.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Verum tVNS (Active Treatment) (Experimental): Participants randomized to receive active transcutaneous auricular vagus nerve stimulation (tVNS) using the Soterix device. Stimulation is delivered nightly for 20 minutes at 80% of the participant's discomfort threshold.
  Interventions: Device: Soterix tVNS device; Behavioral: Sleep Quality; Behavioral: Neurocognitive and mental health outcomes
- Sham tVNS (Placebo Comparator) (Sham Comparator): Participants randomized to receive sham stimulation using the same Soterix device, but with no active electrical stimulation. The procedure mimics the verum condition in duration and setup.
  Interventions: Device: Soterix tVNS device (sham programmed); Behavioral: Sleep Quality; Behavioral: Neurocognitive and mental health outcomes

INTERVENTIONS:
Device: Soterix tVNS device — Active transcutaneous auricular vagus nerve stimulation (tVNS) using the Soterix device.
  Stimulation is delivered nightly for 20 minutes at 80% of the participant's discomfort threshold.
  Other Names: tVNS
  Arms: Verum tVNS (Active Treatment)
Device: Soterix tVNS device (sham programmed) — The sham stimulation used the Soterix device, but without active electrical stimulation. The procedure mimics the verum condition in duration and setup. Inactive stimulation is delivered nightly for 20 minutes at 80% of the participant's discomfort threshold.
  Arms: Sham tVNS (Placebo Comparator)
Behavioral: Sleep Quality — Receive Pittsburgh Sleep Quality Index (PSQI); Insomnia Severity Index (ISI); Sleep diaries; Actigraphy via Fitbit Charge 5
Behavioral: Neurocognitive and mental health outcomes — Measured using CNS Vital Signs and DASS-21.

SUMMARY:
This pilot study will assess the usefulness and potential effectiveness of using transcutaneous auricular vagus nerve stimulation (tVNS) for treating insomnia in adult survivors of childhood acute lymphoblastic leukemia (ALL). Participants will be randomized to receive either active (verum) or inactive (sham) nightly stimulation using a non-invasive earbud device over two time periods: 2 weeks and 8 weeks. The study will assess adherence to the intervention and estimate its effects on sleep quality, stress, and neurocognitive function.

Primary Objective:

Aim 1: To determine a) short-term and b) long-term feasibility of tVNS in terms of participation in ALL Survivors with moderate to severe insomnia.

Aim 2: To estimate the effect size of tVNS on sleep quality, stress, and neurocognitive outcomes in ALL survivors with insomnia.

Exploratory Objectives

Aim 1: To investigate the onset of tVNS effect via actigraphy measures over the intervention epoch.

Aim 2: To estimate the effect size of genetic variants on sleep quality within verum tVNS.

DETAILED DESCRIPTION:
Approximately 40 adult survivors of childhood ALL enrolled in the SJLIFE cohort will be recruited. Eligible participants must have moderate to severe insomnia (ISI ≥8). The intervention involves nightly use of a tVNS device for 20 minutes before sleep. Participants will be randomized to receive either active or sham stimulation. Feasibility will be assessed based on adherence rates, and efficacy will be estimated using subjective (PSQI, ISI) and objective (actigraphy, CNS Vital Signs) measures. Exploratory analyses will examine the onset of tVNS effects and the influence of genetic variants (BDNF rs6265, COMT rs4680) on treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Survivor of Acute Lymphoblastic Leukemia (ALL)
* Enrolled on SJLIFE
* Participant was less than 21 years of age at time of diagnosis.
* Age 20-50 years at the time of enrollment
* Insomnia Severity Index >=8 (Proxy >=8) confirmed prior to enrollment
* Access to home Wi-Fi and Smartphone
* Participant is able to speak and understand the English language
* Participant is able and willing to give consent

Exclusion Criteria:

* Unable to understand the details and requirements of the study (at the discretion of the PI)
* Female participants who are pregnant or planning to become pregnant
* Presence of implanted electrical medical devices (i.e. pacemaker)
* Currently taking medication intended to treat neurocognitive impairment (i.e. stimulants) or medications prescribed for seizure management
* History of skin irritation or other issues during stimulation of inner ear
* Currently utilizing a technological intervention for a sleep disorder (e.g. CPAP)
* Medications and behavioral practices (white noise, night-time yoga, etc) are acceptable as long as the insomnia is persistent.
* History of a contraindicated health condition including:
* Syncope (CTCAE >2)
* Cardiac dysrhythmia (CTCAE >2)
* Vascular Disease (CTCAE >2)
* Coronary Artery Disease (CTCAE >2)
* Active contraindicated heath condition including:
* Cranial Nerve Disorder (CTCAE >2)
* Neuropathy (Cranial Nerves) (CTCAE >2)
* Neuralgia (Cranial Nerves) (CTCAE >2)
* Overt Cerebrovascular Accident (CTCAE >2)
* Seizures (Any in most recent 1 year
* Currently enrolled or participating in any other neurostimulation or neuromodulation ancillary research studies

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Subjective Sleep Quality | Baseline, 2-weeks, 8-weeks
  Pittsburgh Sleep Quality Index (PSQI, 0-57 points). Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported.
Mean change in clinical insomnia score | Baseline, 2-weeks, 8-weeks
  Insomnia Severity Index (ISI, 0-28 points). Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported.
Occurrence of side effects | Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7
  Patient Report of Incidence of Side Effects (PRISE). Descriptive statistics of the change between baseline and 2 and 8 weeks will be reported.
Adherence to intervention | 2-weeks, 8-weeks
  Number of tVNS sessions performed. Descriptive statistics of adherence at 2 weeks and 8 weeks will be reported.
Mean change in Processing Speed (age adjusted z-score) | Baseline, 2-Weeks, 8-weeks
  Symbol Digit Coding Test as the difference between correct responses and errors. Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported.
Mean change in Executive Function (age adjusted z-score) | Baseline, 2-Weeks, 8-weeks
  Shifting Attention Task as the difference between correct responses and errors. Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported.
Mean change in Simple Attention (age adjusted z-score) | Baseline, 2-Weeks, 8-weeks
  Continuous Performance Test as the difference between correct responses and commission errors. Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported.
Mean change in Reaction Time (age adjusted z-score) | Baseline, 2-Weeks, 8-weeks
  Stroop Test as the average of reaction times in the complex and default trials. Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported.
Mean change in Sustained Attention (age adjusted z-score) | Baseline, 2-Weeks, 8-weeks
  Four-Part Continuous Performance Test as the difference between correct responses and incorrect responses in Part 2, 3, and 4. Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported.
Mean change in Working Memory (age adjusted z-score) | Baseline, 2-Weeks, 8-weeks
  Four-Part Continuous Performance Test as the difference between correct responses and incorrect responses in Part 4 only. Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported.
Mean change in Complex Attention (age adjusted z-score) | Baseline, 2-Weeks, 8-weeks
  Evaluated with the Stroop Test (ST), Shifting Attention Test (SAT), and Continuous Performance Test (CPT) as the sum of ST commission errors, SAT errors, CPT commission errors, and CPT omission errors. Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported.
Mean change in Cognitive Flexibility (age adjusted z-score) | Baseline, 2-Weeks, 8-weeks
  Evaluated with the Stroop Test (ST) and Shifting Attention Test (SAT) as the difference between SAT correct responses and the sum of the SAT errors and ST commission errors. Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported.
Mean change in Depression, Anxiety, and Stress (scales) | Baseline, 2-Weeks, 8-weeks
  Evaluated with Depression Anxiety Stress Scale Short Form (DASS SF-21). Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported. DASS SF-21 are reported as population z-scores and categorized into five severity ranges: normal, mild, moderately severe, and extremely severe. The severity levels, higher percentiles being more severe, are determined by z-scores from the DASS manual.
Mean Change in Heart Rate Variability (ms) | Weekly means of daily measurements at baseline, at 2-weeks, and at 8-weeks
  Root Mean Square Successive Difference (RMSSD) of heart rate variability. Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported.
Mean Change in Sleep Onset Latency (minutes) | Weekly means of daily measurements at baseline, at 2-weeks, and at 8-weeks
  Sleep Onset Latency (time in bed before sleep). Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported.
Mean Change in Waking Events (count) | Weekly means of daily measurements at baseline, at 2-weeks, and at 8-weeks
  Number of Awakenings. Descriptive statistics of the difference between experiment arms of the change between baseline and 2 weeks, and baseline and 8 weeks will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Justin E Tanner, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org